CLINICAL TRIAL: NCT00210002
Title: Evaluation of Systematic Intravenous Iron Supplementation During Darbepoetin Alfa Treatment in Prophylaxis of Severe Anaemia Chemo-Induced.
Brief Title: Evaluation of Iron Supplementation During Darbepoetin Alfa Treatment in Prophylaxis of Severe Anaemia Chemo-Induced
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 03 DIVE 01
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-11

CONDITIONS: Neoplasms; Anemia
Keywords: Neoplasms; Solid; Anemia; darbepoetin alfa; ferric saccharose; Venofer®; Aranesp®
MeSH Terms: conditions — Neoplasms; Anemia | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa (Aranesp®)
Drug: Ferric saccharose(Venofer®)

SUMMARY:
The purpose of this study is to evaluate the response rate obtained in an heterogeneous oncologic population treated by chemotherapy, and either by Darbepoetin alfa classic treatment or by association of Darbepoetin alfa -ferric saccharose systematic supplementation, administered concomitantly with chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Well-informed written consent, signed by the patient
* Patient picked up for solid tumor treatment, whichever the localization, with or without metastasis
* Patient revealing, before or during chemotherapy, a moderate anemia, that means: Men: 9<Hb<12 g/dl; Women: 9<Hb<11 g/dl.
* Patient for who at least four chemotherapy cycles are planed (eight in case of weekly chemotherapy) after inclusion in the study
* Patients with life expectancy higher than three months
* Patient with general conditions compatible with the study's follow-up

Exclusion Criteria:

* Contra-indication for Venofer
* Anemia which can have curative treatment
* Bloody transfusion during the previous four weeks
* Documented or suspected medullary invasion
* Uncontrolled arterial hypertension
* Acute bacterial infection
* Transferrin saturation's coefficient
* Pregnancy
* Ferric salts oral treatment interrupted since less than one week
* Patient with bad french language's comprehension
* Patient with a major psychiatric pathology
* Patient under guardianship, trusteeship or justice safeguard

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55
Dates: Start 2003-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Biological response rate for each group.

SECONDARY OUTCOMES:
To determine tolerance for ferric saccharose (Venofer®)
To determine percentage of patients who necessitate an increase of Darbepoetin alfa's dose(Aranesp®)
To determine percentage of hemoglobin rate's correction
To determine biological parameters's evolution

CONTACTS AND LOCATIONS:
Overall Officials: Roland Dugat, Pr, Principal Investigator — Institut Claudius Regaud
Locations (4):
- France (4):
  - Centre Hospitalier de Castres, Castres
  - Centre Hospitalier de Montauban, Montauban
  - Centre Hospitalier Joseph Ducuing, Toulouse
  - Institut Claudius Regaud, Toulouse